CLINICAL TRIAL: NCT03288116
Title: Literature in Mansoura Ophthalmic Center ,Mansoura University
Brief Title: Objective and Subjective Diagnostic Parameters in the Fellow Eye of Unilateral Keratoconus
Status: Completed | Type: Observational
Sponsor: Dar Al Shifa Hospital (Other)
Responsible Party: Principal Investigator, magda torky, clinical professor, Dar Al Shifa Hospital
Other Study IDs: 2352
Record Dates: First submitted 2017-08-30; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patient: Scheimplug imaging and contrast and sensitivity test
  Interventions: Diagnostic Test: Scheimplug imaging and contrast and sensitivity test
- early disease: Scheimplug imaging and contrast and sensitivity test
  Interventions: Diagnostic Test: Scheimplug imaging and contrast and sensitivity test
- normal: Scheimplug imaging and contrast and sensitivity test
  Interventions: Diagnostic Test: Scheimplug imaging and contrast and sensitivity test

INTERVENTIONS:
Diagnostic Test: Scheimplug imaging and contrast and sensitivity test — examination of the patients using the schemiplug imaging with evaluation of keratometric parametres ,pachymetric parametres ,elevation parameters.

SUMMARY:
patients with keratoconus in one eye and forme fruste keratoconus in the fellow eye compared to normal subjects .the patients were examined by schemipflug imaging system (Pentacam)

DETAILED DESCRIPTION:
This cross-sectional study was carried out on patients presenting keratoconus in one eye and forme fruste keratoconus in the fellow eye; the patients attended the outpatient clinic of Mansoura ophthalmic center between January 2014 and February 2015. This study was approved by the institutional research board of the Mansoura faculty of medicine and was performed in accordance with the ethical standards of the Declaration of Helsinki. All patients included in the study provided informed consent.

Ocular examinations were performed on all eyes included in the study. Clinical Keratoconus was diagnosed if all the following criteria were found:1)asymmetric bow tie with skewed radial axis (SRAX), inferior or central steepening on the topography map, 2)mean keratometry (K)>47diopters or an inferior-superior (I-S) value >1.4diopters according to the Rabinowitz and McDonnell criteria[8],and 3)at least one clinical symptom(i.e., stromal thinning, conical protrusion of corneal apex,Fleischer ring, Vogt striae or anterior stromal scar). Forme fruste keratoconus was diagnosed if all the following criteria were found: 1) normal topography, 2) mean K<47D and I-S ≤1.4,3) normal slit lamp, and 4)keratoconus in the fellow eye.

The eyes with an evident keratoconus diagnosis were included in (Group A)and the fellow eyes were included in (Group B).Control cases(Group C) were selected from the normal database of candidates for refractive surgery with the following:1)normal topography, 2)negative rotating Scheimpflug device indices and negative topographic keratoconus classification, 3)normal slit lamp examination, and 4)no history of eye disease(only one eye of each normal candidate was included in the study depending on a computer-based randomizing program).

The exclusion criteria included previous ocular surgery or trauma, significant corneal scarring or associated ocular pathology.

All eyes were examined by rotating Scheimpflug corneal tomography (Pentacam, Oculus Optikgerate GmbH).No patients in the study wore contact lenses. During the Scheimpflug corneal tomography examination, the patient was properly positioned on the chin rest and forehead strap. The patient was asked to blink several times then open both eyes and stare at a fixed target. After obtaining proper alignment, the automatic release mode started the scan; a total of25 single Scheimpflug images were captured within 2 sec for each eye. Three consecutive scans were taken of each eye by the same examiner. The average of the results of three acceptable measurements was included in the study. Each eye was required to have a corneal map with at least 9 mm of corneal coverage and no extrapolated data.

The Pentacam maps were analyzed. The following anterior and posterior corneal surface parameters were evaluated by the Scheimpflug system: corneal dioptric power at the flattest meridian in the 3 mm-central zone(K1),corneal dioptric power in the steepest meridian in the 3mm-central zone (K2)and mean corneal power in the 3mm-zone (mean K).

The pachymetric map was analyzed, including the central corneal thickness (CCT) at the apex of the geometric center and corneal thickness at the thinnest point (CTmin).The average progression index (PPI avg) was calculated as the progression value at the different rings referenced to the mean curve. The minimum (PPI min) and maximum (PPI max) progression indices were recorded. The Ambrósior elational thickness (ART)was calculated as follows: ARTavg=CTmin/PPIavg,ARTmin = CTmin/PPImin, ARTmax =CTmin/PPImax[9].

The posterior corneal elevation maps were evaluated; a reference best fit sphere was calculated at a fixed optical zone of 8 mm, and the posterior corneal elevation values relative to this reference were recorded. The back difference elevation and multimetric D index values were extrapolated from the difference map of the Belin/Ambrósio-enhanced ectasia display of the Pentacam system.

Contrast and Glare sensitivity test:

The contract and glare tests were carried out with a Mesotest II (Oculus Optikgeräte GmbH, Wetzlar, Germany), which consists of Landolt rings of different contrast levels presented in front of a low-brightness background. There are 4 contrast levels, 1:23, 1:5, 1:2.7, and 1:2, which represent the ratio between the light intensity of the optotypes and the background. There were 8 tests, 4 without glare and 4 with glare. Test 1, with a contrast level of 1:23, is the most easily recognized. For statistical purposes, each level of the contrast or glare test was given a score ranging from 20% at the 1:23 level to 100% at the 1:2 level.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically evident keratoconus in one eye and apparently normal in the fellow eye

Exclusion Criteria:

* previous ocular surgery or truama,significant corneal scarring or associatedocular pathology

Ages: 14 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: unilateral keratoconus
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

PRIMARY OUTCOMES:
keratometric power of the corneal surface | 1 year
  in diopter
corneal thickness(pachymetry) | 1 year
  in micrometer
corneal elevations | 1 year
  in micrometer

IPD SHARING:
Plan to Share IPD: No